CLINICAL TRIAL: NCT00527371
Title: Prospective Controlled Trial Comparing Photoselective Vaporization of the Prostate (PVP-120W) to Transurethral Resection of the Prostate (TURP) for the Treatment of Benign Hyperplasia of the Prostate (BPH)
Brief Title: PVP Compared to TURP for the Treatment of Benign Hyperplasia of the Prostate
Acronym: PVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Jean-Eric Tarride, PI, St. Joseph's Healthcare Hamilton
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA 010-0706-01
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign hyperplasia of the prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVP (Experimental): Photoselective vaporization of the prostate.
  Interventions: Device: GreenLight HPS (TM)laser system [Photoselective Vaporization of the prostate (PVP)]
- TURP (Active Comparator): Transurethral resection of the prostate.
  Interventions: Procedure: Transurethral resection of the prostate

INTERVENTIONS:
Device: GreenLight HPS (TM)laser system [Photoselective Vaporization of the prostate (PVP)] — Photoselective vaporization of the prostate will be performed using the GreenLight HPS (TM)laser system (American Medical Systems), which is a high-power (120W) potassium titanyl phosphate (KTP) laser which was licensed by Health Canada in April 2007.
  Other Names: PVP
  Arms: PVP
Procedure: Transurethral resection of the prostate — Transurethral resection of the prostate will be performed with a continuous flow resectoscope and unipolar cautery using a standard technique.
  Other Names: TURP
  Arms: TURP

SUMMARY:
In patients with an enlarged prostate (benign prostatic hyperplasia), is treatment using photoselective vaporization of the prostate (PVP 120 Watt) as effective and cost-effective as the standard treatment of transurethral resection of the prostate (TURP)? A higher-power (120W) laser system has recently been approved by Health Canada for the treatment of an enlarged prostate. This system, which uses laser energy to vaporize the prostate tissue, will be compared with the current standard treatment of transurethral resection of the prostate. This newer generation laser may offer more efficient removal of prostate tissue with fewer complications and may result in clinical and economic benefits compared to the standard treatment. However, there have been no studies comparing the 120W laser with the standard transurethral resection of the prostate. This study will provide currently unavailable information for clinicians and decision makers.

DETAILED DESCRIPTION:
Following a review of treatments for benign prostatic hyperplasia (BPH) by the Medical Advisory Secretariat (MAS) of the Ontario Ministry of Health and Long-Term Care (MOHLTC), the Ontario Health Technology Advisory Committee (OHTAC) recommended that "a registry study be conducted to establish longer term effectiveness and complication rates for PVP given the likelihood of increasing diffusion of this technology". Since then, the Medical Devices Bureau of the Therapeutic Products Directorate, Health Canada, has licensed in April 30, 2007, a 120W-KTP laser system (Greenlight HPS (TM)) for sale in Canada. As several new 120W systems will be operating in Ontario in the coming months, there is an urgent need to evaluate the effectiveness, cost-effectiveness and durability of 120W PVP compared to conventional TURP in the treatment of patients with BPH.

ELIGIBILITY:
Inclusion Criteria:

* Male over the age of 40
* Diagnosed with symptomatic/obstructive symptoms secondary to BPH requiring surgical intervention as determined by their urologist
* Experienced lower urinary tract symptoms (LUTS) secondary to BPH > 3 months in duration
* IPSS value of > 12
* Peak urinary flow < 15mL/sec on voided volume (minimum of 150 ml)
* Prostate size, as measured by transrectal ultrasonography (TRUS), less than 100cc in volume
* American Society of Anesthesiology (ASA) classification of physical status, class 1-3
* Able to read, understand, and sign the Informed Consent
* Willing and able to comply with all follow-up requirements including multiple follow-up visits

Exclusion Criteria:

* Transvesically measured post-void residual volume >400 mL
* Currently in urinary retention
* Chronic urinary retention
* Medications impairing bladder contractibility
* Uncorrectable bleeding disorders or long- term anticoagulation that cannot be stopped
* Recent myocardial infarction or coronary artery stent placement
* Any of the following diseases which appear to involve the bladder: myasthenia gravis, diabetes neuropathy, multiple sclerosis, spinal cord injury or Parkinson disease
* Any patient with idiopathic atonic bladder
* Major pelvic fractures that involved damage to the external urinary sphincter
* Recently completed definitive radiation therapy for prostate cancer
* Active localized or systemic infections; including active urinary tract infection
* Active cystolithiasis, urethral strictures, bladder neck contracture, or acute prostatitis affecting bladder function
* If patient's PSA value > PSA age-adjusted normal value, patient needs to have a negative biopsy before participating in the study
* Confirmed malignancy of the prostate
* Bladder cancer treated with transurethral resection of bladder cancer (TURBT) within 12 months or any patients treated with Bacillius Calmette-Guerin (BCG)
* Bilateral hydronephrosis on renal ultrasound
* Urethral strictures or a residual volume >400 ml
* Immunocompromised
* Previous TURP

Min Age: 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-01; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in International Prostatic Symptom Score (IPSS). | 6-months after surgery versus baseline.

SECONDARY OUTCOMES:
International Prostatic Symptom Score (IPSS) | 1, 3, 12 and 24 months post procedure
Peak or maximum urinary flow rate | 1, 3 and 6 months post surgery
Post-void residual volume | 1, 3, 6 month post procedure
Length of operation/procedure | During procedure
Frequency of blood transfusion | During procedure
Change in hemoglobin in recovery room | Following procedure
Postoperative serum electrolytes (sodium, creatinine) in recovery room | Following procedure
Duration of catheterization | 10 days after procedure
Occurrence of urethral stricture or bladder neck contracture requiring re-operation | up to 2 years after the procedure
Re-bleed rate requiring hospitalization | 1 month after procedure
Prostate-specific antigen (PSA) value | 3 months follow-up
Rate of re-operation | At 1, 6, 12 and 24 months following intervention
Rate of re-catheterization | 1, 6, 12 and 24 months following intervention
Rate of sexual dysfunction (SHIM) and/or retrograde ejaculation (specific question) | Pre-op, 1, 3, 6 months
Use of medications for the treatment of bladder outlet obstruction | 1, 3 and 6 months after intervention
Long-term durability of PVP and TURP (i.e. readmission, drug therapy) | At 12 and 24 months after intervention
IPSS quality of life score (Bother-score) | Pre-op, 1, 3, 6, 12 and 24 months
EQ-5D utility score | Pre-op, 1, 3, 6, 12 and 24 months
Resource utilization: hospital length of stay, OR time, pain medications, follow-up care (e.g. urologist visits, lab tests) | Pre-op, 1, 3, 6, 12 and 24 months
Productivity losses | Pre-op, 1, 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Eric Tarride, PhD, Study Chair — Program for Assessment of Technology in Health, St. Joseph's Healthcare/McMaster University; Gary McIsaac, MD, Principal Investigator — Trillium Health Centre; Edward Woods, MD, Principal Investigator — The Scarborough Hospital; Paul Whelan, MD, Principal Investigator — McMaster Institute of Urology at St. Joseph's Healthcare Hamilton
Locations (3):
- Canada (3):
  - McMaster Institute of Urology at St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - The Scarborough Hospital, Scarborough Village, Ontario

REFERENCES:
- [Result] Whelan JP, Bowen JM, Burke N, Woods EA, McIssac GP, Hopkins RB, O'Reilly DJ, Xie F, Sehatzadeh S, Levin L, Mathew SP, Patterson LL, Goeree R, Tarride JE. A prospective trial of GreenLight PVP (HPS120) versus transurethral resection of the prostate in the treatment of lower urinary tract symptoms in Ontario, Canada. Can Urol Assoc J. 2013 Sep-Oct;7(9-10):335-41. doi: 10.5489/cuaj.180. PMID 24319513
- [Result] Bowen JM, Whelan JP, Hopkins RB, Burke N, Woods EA, McIsaac GP, O'Reilly DJ, Xie F, Sehatzadeh S, Levin L, Mathew SP, Patterson LL, Goeree R, Tarride JE. Photoselective vaporization for the treatment of benign prostatic hyperplasia. Ont Health Technol Assess Ser. 2013 Aug 1;13(2):1-34. eCollection 2013. PMID 24019857